CLINICAL TRIAL: NCT02946918
Title: Levothyroxine Replacement With Liquid Gel Capsules or Tablets in Post-thyroidectomy Stage in Low Risk Differentiated Thyroid Cancer Patients
Brief Title: Levothyroxine Replacement With Liquid Gel Capsules vs Tablets Post-thyroidectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminating study as sponsor has sold the drug to another company
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Akrimax Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Alex Tessnow, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU 022015-044
Record Dates: First submitted 2016-10-21; First posted 2016-10-27 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Thyroid Cancer; Postsurgical Hypothyroidism
Keywords: levothyroxine
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tablets (Experimental): Patients in this arm will receive levothyroxine tablets (encapsulated for blinding purposes)
  Interventions: Drug: Levothyroxine
- Gelcaps (Experimental): Patients in this arm will receive levothyroxine gelcaps (encapsulated for blinding purposes)
  Interventions: Drug: Levothyroxine

INTERVENTIONS:
Drug: Levothyroxine — Patients post-thyroidectomy will receive either levothyroxine in tablet form or in gelcaps. Initial dose 1.5-1.8 mcg per kg, orally and daily
  Other Names: Tirosint, Synthroid

SUMMARY:
In some patients, levothyroxine liquid gel capsules may demonstrate superior absorption than the tablet option. Impaired absorption of thyroid hormone directly correlates to higher and more unpredictable TSH (thyroid stimulating hormone) levels.

The investigators therefore hypothesize that following thyroidectomy for Stage I/II differentiated thyroid cancer the gel capsule levothyroxine formulation will provide more predictable TSH results and in turn require fewer dose adjustments to achieve optimal hormone levels in the postoperative period.

The aim of this investigation is to compare the use of levothyroxine in liquid gel capsules to tablet form for TSH suppression following thyroidectomy for presumed stage I/II differentiated thyroid cancer.

DETAILED DESCRIPTION:
Ten patients will be randomized prior to surgery to receive levothyroxine in tablet form and ten patients will be randomized to receive in gel capsule form. Both forms will be encapsulated in order to allow double-blinding of the study.

The postoperative goal TSH will be between 0.1 and 0.5 mU/L (milli units per litre) in both arms.

Patients will be seen at weeks 6, 12 and 18 postoperatively and have TSH and Free T4 measured. The primary outcome is the number of patients at each visit that are at goal range TSH.

A secondary analysis will compare the dose changes required between the two groups in order to achieve goal TSH.

Another secondary analysis will investigate the patients' quality of life. Two different surveys (see secondary outcomes below) will be performed at both study entry and completion to compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Presumed AJCC (American Joint Committee on Cancer) tumor Stage I or II
* Planned total or near-total thyroidectomy
* Planned goal TSH suppression 0.1-0.5 mU/L for at least 18 weeks postoperatively
* Normal serum TSH within 12 months preceding surgery

Exclusion Criteria:

* AJCC Stage III or greater
* Undifferentiated, Anaplastic or Medullary Thyroid Cancer
* Planned postoperative TSH goal other than 0.1-0.5 mU/L
* History of gastrointestinal malabsorption or gastric bypass surgery
* Pregnancy
* Use of medications that alter the absorption or metabolism of levothyroxine
* Prior use of levothyroxine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Tessnow, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vita R, Fallahi P, Antonelli A, Benvenga S. The administration of L-thyroxine as soft gel capsule or liquid solution. Expert Opin Drug Deliv. 2014 Jul;11(7):1103-11. doi: 10.1517/17425247.2014.918101. Epub 2014 Jun 4. PMID 24896369
- [Background] McMillan CV, Bradley C, Woodcock A, Razvi S, Weaver JU. Design of new questionnaires to measure quality of life and treatment satisfaction in hypothyroidism. Thyroid. 2004 Nov;14(11):916-25. doi: 10.1089/thy.2004.14.916. PMID 15671770

RESULTS

PARTICIPANT FLOW:
Groups:
- Tablets: Patients in this arm will receive levothyroxine tablets (encapsulated for blinding purposes)
  Levothyroxine: Patients post-thyroidectomy will receive either levothyroxine in tablet form or in gelcaps
- Gelcaps: Patients in this arm will receive levothyroxine gelcaps (encapsulated for blinding purposes)
  Levothyroxine: Patients post-thyroidectomy will receive either levothyroxine in tablet form or in gelcaps
Period: Overall Study
Arm/Group | Tablets | Gelcaps
Started | 6 | 8
Completed | 5 | 5
Not Completed | 1 | 3
Not completed — Patient unblinded himself | 1 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Ran out of study medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tablets | Gelcaps | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 7 | 12
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 10
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 7 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each Group at Predefined Target TSH Range at 18 Weeks
Description: The target TSH (Thyroid stimulating hormone) range will be 0.1 to 0.5 mU/L. The number of patients in each arm (gelcaps or tablets) who are in this range at the completion of the study (18 weeks) will be assessed and the data compared at completion of the study.
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tablets | Gelcaps
Number analyzed (Participants) | 6 | 8
Participants | 2 | 4

2. Secondary Outcome: Mean Number of Dose Adjustments
Description: The number of dose adjustments required to attain TSH target range for each formulation will be tabulated and the data compared at the end of the study
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: The number of dose adjustments
Arm/Group | Tablets | Gelcaps
Number analyzed (Participants) | 6 | 8
The number of dose adjustments | 2.0 (0.63) | 1.25 (1.04)

3. Secondary Outcome: Change in Mean Patient Quality of Life Score
Description: Patients will be administered survey (Thyroid-Dependent Quality of Life ) to assess their quality of life (at the beginning of the study and again at study completion). The results of these scores will be tabulated and compared between the two arms. Possible score range from 0 to 450; lower score means improved quality of life.
Time Frame: Baseline,18 weeks
Population: Out of 6 people from the Tablet group, 1 did not complete the second survey. Out of 8 people from the Gelcap group, 3 people did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tablets | Gelcaps
Number analyzed (Participants) | 5 | 5
score on a scale | -1.2 (12.99) | -29.6 (48.06)

4. Secondary Outcome: Treatment Satisfaction Survey
Description: The Thyroid Treatment Satisfaction Questionnaire Measures the treatment satisfaction. Possible measure 0 to 42; Higher the score, better the outcome (more satisfied the patient)
Time Frame: 18 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tablets | Gelcaps
Number analyzed (Participants) | 5 | 5
score on a scale | 39.2 (3.70) | 39 (3)

ADVERSE EVENTS:
Time Frame: 18 weeks (until completion of the study)
Description: All 14 subjects were considered at risk for adverse events
Arm/Group | Tablets | Gelcaps
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 4/6 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tablets (N=6) | Gelcaps (N=8)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
anxiety (Nervous system disorders) | 1 (1) | 1 (1)
psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
fatigue (Endocrine disorders) | 1 (1) | 1 (1)
hypocalcemia (Endocrine disorders) | 1 (1) | 0 (0)
rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT02946918/Prot_SAP_000.pdf